CLINICAL TRIAL: NCT02757287
Title: Desogestrel and Corifollitropin Treatment for Ovarian Stimulation in Donors
Brief Title: Desogestrel (DSG) and Corifollitropin(FSH-CTP) Alfa for Ovarian Stimulation in Donors
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Fundacion Dexeus (Other)
Collaborators: Fundación Dexeus Salud de la Mujer (Unknown)
Responsible Party: Principal Investigator, Dr. Francisca Martínez, PhD, Fundacion Dexeus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMD-DES-2016-01
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Infertility
Keywords: Ovarian stimulation; LH inhibition
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FSH-CTP + DESOGESTREL (Experimental): Single injection of FSH-CTP and oral desogestrel since the first menstruation day, until bolus of GnRH agonist to follicular maturation
  Interventions: Drug: FSH-CTP + DESOGESTREL

INTERVENTIONS:
Drug: FSH-CTP + DESOGESTREL — Hormones measured on day of 7th menstrual cycle day , day of pre-ovulatory bolus of GnRH and the day after the bolus ( estradiol, FSH, Progesterone, LH)
  - Quality of Life questionnaire the day after the bolus

SUMMARY:
Currently, controlled ovarian stimulation (COS) in oocyte donors is performed by daily injections of gonadotropins( recombinant FSH) plus a GnRH Antagonist usually form 5th-6th stimulation day until ovulation induction with a bolus of another injection of a gonadotropin-releasing hormone (GnRH) Agonist. Injections of the GnRH Antagonist avoid untimely luteinizing hormone (LH) surge and spontaneous ovulation prior to follicular aspiration. There is a preparation of long-acting recombinant follicle stimulating hormone (rFSH= (corifollitropin alfa (FSH-CTP), Elonva®, MSD), that allows that a single subcutaneous injection substitutes the first 7 days of daily gonadotropin injections. On the other hand, a contraceptive oral progesterone only( Desogestrel, DSG) is available for contraception, avoiding the LH surge. It has been described the usefulness of orally administered medroxyprogesterone acetate, 10 mg to inhibit the endogenous LH surge in IVF patients during COS.

In donors, by administering a single injection of FSH-CTP and oral desogestrel since the first menstruation day, the total number of injections administered is reduced and less discomfort is experienced without adverse impact on ovarian response. No description of the hormonal and ovarian response under this protocol has been published

DETAILED DESCRIPTION:
* oral desogestrel since the first menstruation day,
* a single injection of FSH-CTP on the 7th menstrual cycle day
* routine monitoring of ovarian response with transvaginal ultrasound every second day until pre-ovulatory bolus of GnRH
* Hormones measured on day of 7th menstrual cycle day , day of pre-ovulatory bolus of GnRH and the day after the bolus ( estradiol, FSH, Progesterone, LH)
* Quality of Life questionnaire the day after the bolus

ELIGIBILITY:
Inclusion Criteria:

* Population: donors (18-35 ) from candidates of Donor program
* Fulfilling inclusión medical and legal criteria (RD -Ley de transposición de la normativa europea a la legislación española 9/2014)
* Who had had undergone previously convencional COS (controlled ovarian stimulation) with FSH-CTP and daily antagonist injections
* Given signed consent form.

Exclusion Criteria:

* Previous low response to COS
* Previous ovarian hyperstimulation syndrome.
* Ovarian cysts.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Total dose of gonadotrophins | At the end of the stimulation treatment period (5 or 7 days after begining of treatment)
  Total Consume of gonadotrophins

SECONDARY OUTCOMES:
Plasma LH | Day of GnrH bolus
  Level of LH in plasma (mIU/ml)
Number of mature oocytes | Day of oocyte recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Quiron Dexeus, Barcelona, Spain

REFERENCES:
- [Background] Martinez F, Boada M, Coroleu B, Clua E, Parera N, Rodriguez I, Barri PN. A prospective trial comparing oocyte donor ovarian response and recipient pregnancy rates between suppression with gonadotrophin-releasing hormone agonist (GnRHa) alone and dual suppression with a contraceptive vaginal ring and GnRH. Hum Reprod. 2006 Aug;21(8):2121-5. doi: 10.1093/humrep/del121. Epub 2006 Apr 21. PMID 16632462
- [Background] Martinez F, Clua E, Santmarti P, Boada M, Rodriguez I, Coroleu B. Randomized, comparative pilot study of pituitary suppression with depot leuprorelin versus cetrorelix acetate 3 mg in gonadotropin stimulation protocols for oocyte donors. Fertil Steril. 2010 Nov;94(6):2433-6. doi: 10.1016/j.fertnstert.2010.02.059. Epub 2010 Apr 28. PMID 20430379
- [Background] Requena A, Cruz M, Collado D, Izquierdo A, Ballesteros A, Munoz M, Garcia-Velasco JA. Evaluation of the degree of satisfaction in oocyte donors using sustained-release FSH corifollitropin alpha. Reprod Biomed Online. 2013 Mar;26(3):253-9. doi: 10.1016/j.rbmo.2012.11.015. Epub 2012 Dec 5. PMID 23352098
- See also: Related Info — http://www.dexeus.com/